CLINICAL TRIAL: NCT03355053
Title: Investigation of Sleep in the Intensive Care Unit
Acronym: ICU-SLEEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Michael Brandon Westover, MD/PhD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017P000090; R01NS102190 (NIH)
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Delirium; Sleep
MeSH Terms: conditions — Delirium | interventions — Dexmedetomidine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, phase II, double-blind, placebo-controlled, three-arm, parallel-group, mechanistic, randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dexmedetomidine, continuous very-low-dose overnight infusion (Active Comparator): Patients randomized to this study arm will receive dexmedetomidine, given as a very-low-dose (0.1 mcg/kg/hour group; rate of 0.075 mL/kg/hour at a concentration of 1.33 mcg/mL) continuous overnight infusion. Study drug will be provided by the MGH research pharmacy as a clear liquid and delivered by the research staff directly to the patient's ICU nurse, in a 60 mL syringe/bag (s). Nursing will then administer the study drug intravenously each night (11 hours; 8PM through 7AM) until either discharge from the ICU or up to 7 consecutive nights, whichever occurs first.
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine, continuous low-dose overnight infusion (Active Comparator): Patients randomized to this study arm will receive dexmedetomidine, given as a low-dose (0.3 mcg/kg/hour group; rate of 0.075 mL/kg/hour at a concentration of 4 mcg/mL) continuous overnight infusion. Study drug will be provided by the MGH research pharmacy as a clear liquid and delivered by the research staff directly to the patient's ICU nurse, in a 60 mL syringe/bag (s). Nursing will then administer the study drug intravenously each night (11 hours; 8PM through 7AM) until either discharge from the ICU or up to 7 consecutive nights, whichever occurs first.
  Interventions: Drug: Dexmedetomidine
- Usual care and placebo (normal saline) (Placebo Comparator): Patients randomized to this study arm will receive standard ICU care plus a normal saline placebo, given as a continuous overnight infusion, at a rate of 0.075 mL/kg/hour. Study drug will be provided by the MGH research pharmacy as a clear liquid and delivered by the research staff directly to the patient's ICU nurse, in a 60 mL syringe/bag (s). Nursing will then administer the study drug intravenously each night (11 hours; 8PM through 7AM) until either discharge from the ICU or up to 7 consecutive nights, whichever occurs first.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — "Dex (Precedex, Dexmedetomidine HCl Injection) is produced by Pfizer Inc, NY, Ny (formerly Hospira). Dex is a white or almost white powder that is freely soluble in water and has a pKa of 7.1. Its partition coefficient in-octanol: water at pH 7.4 is 2.89. Dex is supplied as a clear, colorless, isotonic solution with a pH of 4.5 to 7.0. Each mL contains 118 mcg of dexmedetomidine hydrochloride equivalent to 100 mcg (0.1mg) of dexmedetomidine and 9 mg of sodium chloride in water. The solution is preservative-free and contains no additives or chemical stabilizers. The MGH Pharmacy currently obtains Dex from the supplier as a solution in 50 mL clear-glass bottles, as a clear liquid, at a concentration of 4mcg/mL."
  Other Names: Precedex (dexmedetomidine hydrochloride; Pfizer Inc, NY, Ny)
  Arms: Dexmedetomidine, continuous low-dose overnight infusion; Dexmedetomidine, continuous very-low-dose overnight infusion
Drug: Placebo — From the package insert: "0.9% Sodium Chloride Injection, USP is sterile and nonpyrogenic. It is produced by Pfizer Inc, NY, Ny (formerly Hospira). It is a parenteral solution containing sodium chloride in water for injection intended for intravenous administration. Each 100 mL of 0.9% Sodium Chloride Injection, USP contains 900 mg sodium chloride in water for injection. Electrolytes per 1000 mL: sodium (Na+ ) 154 mEq; chloride (Cl- ) 154 mEq. The osmolarity is 308 mOsmol/L (calc.). The pH is 5.6 (4.5 to 7.0). This solution contains no bacteriostat, antimicrobial agent or added buffer and is intended only as a single-dose injection. When smaller doses are required, the unused portion should be discarded. 0.9% Sodium Chloride Injection, USP is a parenteral fluid and electrolyte replenisher. Sodium Chloride, USP is chemically designated NaCl, a white crystalline powder freely soluble in water. Water for Injection, USP is chemically designated H2O."
  Other Names: Normal saline (0.9% Sodium Chloride; Pfizer Inc, NY, Ny)
  Arms: Usual care and placebo (normal saline)

SUMMARY:
Sleep deprivation is common and often severe in critically ill patients cared for in intensive care units (ICUs) and is hypothesized to be a modifiable risk factor for delirium, which in turn is hypothesized to be a modifiable risk factor for long-term cognitive disability following recovery from critical illness. Dexmedetomidine (Dex) reduces the incidence of delirium in ICU patients by unknown mechanisms. The Investigation of Sleep in the Intensive Care Unit (ICU-SLEEP) Trial aims to determine whether Dex reduces delirium by improving sleep, whether a low- and/or very-low dose continuous infusion of Dex increases delirium-free days more, and the relationship between sleep deprivation in the ICU to long-term cognitive outcomes.

DETAILED DESCRIPTION:
Sleep deprivation is among the most common complaints about the ICU experience. ICU sleep tends to be light and non-restorative (as opposed to deep/restorative sleep), severely fragmented, and distributed throughout the day and night rather than consolidated into nighttime hours. Sleep-deprived patients suffer from sleep debt, a condition of impaired attention and memory, and cognitive slowing. Sleep disturbances in the ICU arise not only from light and noise pollution, but also from drugs that interfere with brain activity involved in restorative sleep. Sleep deprivation has also been suggested as a major modifiable risk factor for acute encephalopathy, also known as delirium. Delirium is an acute state of confusion that affects up to 50% of non-ventilated ICU patients and is one of six leading causes of preventable morbidity and mortality in hospitalized elderly patients. Many patients who survive delirium experience long-term cognitive impairment and loss of independence. Current medications used in the ICU to treat sleep problems (e.g. benzodiazepines, antipsychotics) do not induce natural sleep and do not prevent delirium. In contrast, the investigators have found that the α2-adrenoceptor agonist dexmedetomidine can induce biomimetic sleep, a brain state whose pattern of electroencephalogram (EEG) activity, cerebral blood flow, and functional connectivity approximates restorative sleep. Moreover, a recent large clinical trial in post-surgical patients suggests that low-dose dexmedetomidine given overnight substantially reduces the risk of delirium. It is unknown whether this benefit is linked to improved sleep, or whether patients with better sleep while in the ICU have better long-term cognitive outcomes. The investigator's central hypothesis is that sleep deprivation substantially mediates both the short- and long-term cognitive impairments associated with delirium in critical illness. To test this hypothesis, the ICU-SLEEP trial aims to: 1A) Compare the burden of delirium, as measured by the number of delirium-free days (DFDs), in ICU patients non-ventilated at study enrollment, who are receiving biomimetic sleep induced by Dex, given as a continuous overnight 1) very-low-dose or 2) low-dose infusion vs. 3) usual care and placebo; 1B) Assess whether the 1) very-low-dose continuous overnight infusion of Dex increases DFDs compared to the 2) low-dose continuous overnight infusion; 2A) Determine whether Dex reduces ICU delirium via reducing sleep deprivation, using causal mediation analysis; 2B) Determine the associations between specific components of acute cognitive impairment, seen in sleep deprivation and delirium, with specific measures of sleep deprivation; 3A) Determine whether ICU patients treated with Dex while in the hospital have a lower incidence of long-term cognitive impairment; 3B) Determine whether any differences in long-term cognitive impairment between ICU survivors treated with Dex vs. usual care and placebo are mediated by differences in sleep deprivation. The knowledge gained will provide insights into the mechanisms by which Dex prevents delirium and guidance on the optimal dosing strategy for prophylactic Dex, which can be used to design pivotal phase 3 clinical trials.

ELIGIBILITY:
Inclusion Criteria

1. Admitted or scheduled to be admitted to an MGH medical or surgical ICU (Blake 7 or 12, or Ellison 4)
2. Male or female, aged ≥ 50 years
3. Provision of signed and dated informed consent form (by patient or legally authorized representative (LAR))
4. Stated willingness to comply with all study procedures and availability for the duration of the study
5. Not on mechanical ventilation at the time of enrollment
6. Able to be enrolled before 7PM
7. For females of reproductive potential: pregnancy test is negative

Exclusion Criteria

1. Dementia, as measured by a score of ≥3.3 on the Informant Questionnaire on Cognitive Decline in the Elderly Short Form (IQCODE-SF)
2. Unable to be assessed for delirium (e.g. blindness or deafness)
3. Follow-up would be difficult (e.g. active substance abuse, homelessness)
4. Pregnancy or lactation
5. Known pre-existing neurologic disease or injury with focal neurologic or cognitive deficits
6. Serious cardiac disease (e.g. sick sinus syndrome without a pacemaker, sinus bradycardia, second- or third-degree AV block, congestive heart failure with ejection fraction <30%)
7. Severe liver dysfunction (Child-Pugh class C)
8. Severe renal dysfunction (receiving dialysis)
9. Low likelihood of survival >24 hours
10. Low likelihood of staying in ICU overnight
11. Known allergic reactions to components of dexmedetomidine
12. Patient is receiving or planning to go on dexmedetomidine at the time of enrollment
13. Patient is receiving either of the anticholinergic drugs scopolamine or penehyclidine; or alpha-2-agonist clonidine
14. Concomitant enrollment in another study protocol that may interfere with data acquisition or reliability of measurements
15. Deemed unsuitable for selection by the research team or ICU providers due to any medical, legal, social, language (non-English speaking) or interpersonal issues that would either compromise the study or the routine care of patients

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 522 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
In-hospital Delirium-free days (IH-DFDs) | First 14 hospital days from start of infusion [or until hospital discharge, whichever occurs first]
  In-hospital Delirium-free days (IH-DFDs) are calculated as the sum of days without delirium during the first 14 hospital days from start of infusion in the two Dex treatment arms combined (arms 1 and 2) vs. usual care (arm 3). Delirium is defined as any positive Confusion Assessment Method (CAM) or CAM for the ICU (CAM-ICU) assessment, with each yielding a binary result (1 = delirious/CAM+, 0 = non-delirious/CAM-). For each patient, delirium is assessed twice daily. If a patient has any positive delirium assessments on any given day of the assessment days, they are considered to have had delirium during these days. Days with coma are counted together with delirium.

SECONDARY OUTCOMES:
ICU-Delirium-free days (ICU-DFDs) | First 7 ICU days from start of infusion [or until ICU discharge, whichever occurs first]
  ICU-Delirium-free days (ICU-DFDs) are calculated as the sum of days without delirium during the first 7 ICU days from start of infusion in the two Dex treatment arms combined (arms 1 and 2) vs. usual care (arm 3). Delirium is defined as any positive Confusion Assessment Method (CAM) or CAM for the ICU (CAM-ICU) assessment, with each yielding a binary result (1 = delirious/CAM+, 0 = non-delirious/CAM-). For each patient, delirium is assessed twice daily. If a patient has any positive delirium assessments on any given day of the assessment days, they are considered to have had delirium during these days. Days with coma are counted together with delirium.
Sleep Quantity-quality (SQ) score | First 14 ICU days from start of infusion [or until ICU discharge, whichever occurs first]
  The Sleep Quantity-quality (SQ) score is a sleep composite measure formed by averaging the z-scores for raw measures of sleep quality (total sleep time (TST), sleep fragmentation index (SFI), time in N2, time in N3), where a higher SQ score indicates better outcomes.
Acute Cognitive Function (ACF) score | First 14 ICU days from start of infusion [or until ICU discharge, whichever occurs first]
  The Acute Cognitive Function (ACF) score is a reliable change index controlling for practice effects (RCI+PE) for a composite of acute cognitive measures. These include twice daily Confusion Assessment Method-Severity (CAM-S; Short Form (0-7) & Long Form (0-19), where higher scores indicate increased severity of delirium symptoms); and Psychomotor Vigilance Test (PVT) scores collected in the first 7 ICU days from start of infusion [or until ICU discharge, whichever occurs first]. Composites will be formed by averaging z-scores for CAM-S and PVT scores, where a higher ACF score indicates better outcomes.
Long-term Cognitive Function (LCF) score | 3-, 6-, and 12 months post-enrollment
  The Long-term Cognitive Function (LCF) score is a composite average of z-scores from long-term cognitive outcome measures of the different components, where a higher LCF score indicates better outcomes.

OTHER OUTCOMES:
Spearman correlation coefficient (rho) between sleep quality and acute cognitive function | First 14 ICU days from start of infusion [or until ICU discharge, whichever occurs first]
  Spearman's correlation coefficient (rho) describes the correlation between sleep quality on the previous night, as measured by the Sleep Quantity-quality (SQ) score, and acute cognitive function, as measured by the Acute Cognitive Function (ACF) score.
Average Causal Mediation Effect (ACME) of sleep deprivation on delirium-free days | First 14 ICU days from start of infusion [or until ICU discharge, whichever occurs first]
  Causal effect of sleep deprivation (SD) on In-hospital Delirium-free days (IH-DFDs) and ICU-Delirium-free days (ICU-DFDs), where SD is quantified by the Sleep Quantity-quality (SQ) score.
Average Causal Mediation Effect (ACME) of sleep deprivation on acute cognitive outcomes | First 14 ICU days from start of infusion [or until ICU discharge, whichever occurs first]
  Causal effect of sleep deprivation (SD) on acute cognitive outcomes, where SD is quantified by the Sleep Quantity-quality (SQ) score, and acute cognitive function is quantified by the Acute Cognitive Function (ACF) score.
Average Causal Mediation Effect (ACME) of sleep deprivation on long-term cognitive outcomes | First 14 ICU days from start of infusion [or until ICU discharge, whichever occurs first]; 3-, 6-, and 12 months post-enrollment
  Causal effect of sleep deprivation (SD) on long-term cognitive outcomes, where SD is quantified by the Sleep Quantity-quality (SQ) score, and long-term cognitive function is quantified by the Long-term Cognitive Function (LCF) score.

CONTACTS AND LOCATIONS:
Overall Officials: M. Brandon Westover, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hardin KA, Seyal M, Stewart T, Bonekat HW. Sleep in critically ill chemically paralyzed patients requiring mechanical ventilation. Chest. 2006 Jun;129(6):1468-77. doi: 10.1378/chest.129.6.1468. PMID 16778263
- [Background] Fanfulla F, Ceriana P, D'Artavilla Lupo N, Trentin R, Frigerio F, Nava S. Sleep disturbances in patients admitted to a step-down unit after ICU discharge: the role of mechanical ventilation. Sleep. 2011 Mar 1;34(3):355-62. doi: 10.1093/sleep/34.3.355. PMID 21358853
- [Background] Gabor JY, Cooper AB, Hanly PJ. Sleep disruption in the intensive care unit. Curr Opin Crit Care. 2001 Feb;7(1):21-7. doi: 10.1097/00075198-200102000-00004. PMID 11373507
- [Background] Mundigler G, Delle-Karth G, Koreny M, Zehetgruber M, Steindl-Munda P, Marktl W, Ferti L, Siostrzonek P. Impaired circadian rhythm of melatonin secretion in sedated critically ill patients with severe sepsis. Crit Care Med. 2002 Mar;30(3):536-40. doi: 10.1097/00003246-200203000-00007. PMID 11990911
- [Background] Trompeo AC, Vidi Y, Locane MD, Braghiroli A, Mascia L, Bosma K, Ranieri VM. Sleep disturbances in the critically ill patients: role of delirium and sedative agents. Minerva Anestesiol. 2011 Jun;77(6):604-12. PMID 21617624
- [Background] Parthasarathy S, Tobin MJ. Effect of ventilator mode on sleep quality in critically ill patients. Am J Respir Crit Care Med. 2002 Dec 1;166(11):1423-9. doi: 10.1164/rccm.200209-999OC. Epub 2002 Sep 5. PMID 12406837
- [Background] Wilson JE, Mart MF, Cunningham C, Shehabi Y, Girard TD, MacLullich AMJ, Slooter AJC, Ely EW. Delirium. Nat Rev Dis Primers. 2020 Nov 12;6(1):90. doi: 10.1038/s41572-020-00223-4. PMID 33184265
- [Background] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- [Background] Mart MF, Williams Roberson S, Salas B, Pandharipande PP, Ely EW. Prevention and Management of Delirium in the Intensive Care Unit. Semin Respir Crit Care Med. 2021 Feb;42(1):112-126. doi: 10.1055/s-0040-1710572. Epub 2020 Aug 3. PMID 32746469
- [Background] Leslie DL, Marcantonio ER, Zhang Y, Leo-Summers L, Inouye SK. One-year health care costs associated with delirium in the elderly population. Arch Intern Med. 2008 Jan 14;168(1):27-32. doi: 10.1001/archinternmed.2007.4. PMID 18195192
- [Background] Vasilevskis EE, Chandrasekhar R, Holtze CH, Graves J, Speroff T, Girard TD, Patel MB, Hughes CG, Cao A, Pandharipande PP, Ely EW. The Cost of ICU Delirium and Coma in the Intensive Care Unit Patient. Med Care. 2018 Oct;56(10):890-897. doi: 10.1097/MLR.0000000000000975. PMID 30179988
- [Background] Diekelmann S, Born J. The memory function of sleep. Nat Rev Neurosci. 2010 Feb;11(2):114-26. doi: 10.1038/nrn2762. Epub 2010 Jan 4. PMID 20046194
- [Background] Ngo HV, Martinetz T, Born J, Molle M. Auditory closed-loop stimulation of the sleep slow oscillation enhances memory. Neuron. 2013 May 8;78(3):545-53. doi: 10.1016/j.neuron.2013.03.006. Epub 2013 Apr 11. PMID 23583623
- [Background] Staresina BP, Bergmann TO, Bonnefond M, van der Meij R, Jensen O, Deuker L, Elger CE, Axmacher N, Fell J. Hierarchical nesting of slow oscillations, spindles and ripples in the human hippocampus during sleep. Nat Neurosci. 2015 Nov;18(11):1679-1686. doi: 10.1038/nn.4119. Epub 2015 Sep 21. PMID 26389842
- [Background] Nedergaard M. Neuroscience. Garbage truck of the brain. Science. 2013 Jun 28;340(6140):1529-30. doi: 10.1126/science.1240514. PMID 23812703
- [Background] Xie L, Kang H, Xu Q, Chen MJ, Liao Y, Thiyagarajan M, O'Donnell J, Christensen DJ, Nicholson C, Iliff JJ, Takano T, Deane R, Nedergaard M. Sleep drives metabolite clearance from the adult brain. Science. 2013 Oct 18;342(6156):373-7. doi: 10.1126/science.1241224. PMID 24136970
- [Background] Sfera A, Osorio C. Water for thought: is there a role for aquaporin channels in delirium? Front Psychiatry. 2014 May 26;5:57. doi: 10.3389/fpsyt.2014.00057. eCollection 2014. No abstract available. PMID 24904440
- [Background] Sfera A, Osorio C, Price AI, Gradini R, Cummings M. Delirium from the gliocentric perspective. Front Cell Neurosci. 2015 May 11;9:171. doi: 10.3389/fncel.2015.00171. eCollection 2015. PMID 26029046
- [Background] Bondareff W, Mountjoy CQ, Roth M. Selective loss of neurones of origin of adrenergic projection to cerebral cortex (nucleus locus coeruleus) in senile dementia. Lancet. 1981 Apr 4;1(8223):783-4. doi: 10.1016/s0140-6736(81)92657-x. No abstract available. PMID 6110985
- [Background] Haack M, Sanchez E, Mullington JM. Elevated inflammatory markers in response to prolonged sleep restriction are associated with increased pain experience in healthy volunteers. Sleep. 2007 Sep;30(9):1145-52. doi: 10.1093/sleep/30.9.1145. PMID 17910386
- [Background] Munster BC, Aronica E, Zwinderman AH, Eikelenboom P, Cunningham C, Rooij SE. Neuroinflammation in delirium: a postmortem case-control study. Rejuvenation Res. 2011 Dec;14(6):615-22. doi: 10.1089/rej.2011.1185. Epub 2011 Oct 6. PMID 21978081
- [Background] Akeju O, Pavone KJ, Westover MB, Vazquez R, Prerau MJ, Harrell PG, Hartnack KE, Rhee J, Sampson AL, Habeeb K, Gao L, Pierce ET, Walsh JL, Brown EN, Purdon PL. A comparison of propofol- and dexmedetomidine-induced electroencephalogram dynamics using spectral and coherence analysis. Anesthesiology. 2014 Nov;121(5):978-89. doi: 10.1097/ALN.0000000000000419. PMID 25187999
- [Background] Pandharipande P, Shintani A, Peterson J, Pun BT, Wilkinson GR, Dittus RS, Bernard GR, Ely EW. Lorazepam is an independent risk factor for transitioning to delirium in intensive care unit patients. Anesthesiology. 2006 Jan;104(1):21-6. doi: 10.1097/00000542-200601000-00005. PMID 16394685
- [Background] Seymour CW, Pandharipande PP, Koestner T, Hudson LD, Thompson JL, Shintani AK, Ely EW, Girard TD. Diurnal sedative changes during intensive care: impact on liberation from mechanical ventilation and delirium. Crit Care Med. 2012 Oct;40(10):2788-96. doi: 10.1097/CCM.0b013e31825b8ade. PMID 22824928
- [Background] Pandharipande PP, Pun BT, Herr DL, Maze M, Girard TD, Miller RR, Shintani AK, Thompson JL, Jackson JC, Deppen SA, Stiles RA, Dittus RS, Bernard GR, Ely EW. Effect of sedation with dexmedetomidine vs lorazepam on acute brain dysfunction in mechanically ventilated patients: the MENDS randomized controlled trial. JAMA. 2007 Dec 12;298(22):2644-53. doi: 10.1001/jama.298.22.2644. PMID 18073360
- [Background] Maldonado JR, Wysong A, van der Starre PJ, Block T, Miller C, Reitz BA. Dexmedetomidine and the reduction of postoperative delirium after cardiac surgery. Psychosomatics. 2009 May-Jun;50(3):206-17. doi: 10.1176/appi.psy.50.3.206. PMID 19567759
- [Background] Riker RR, Shehabi Y, Bokesch PM, Ceraso D, Wisemandle W, Koura F, Whitten P, Margolis BD, Byrne DW, Ely EW, Rocha MG; SEDCOM (Safety and Efficacy of Dexmedetomidine Compared With Midazolam) Study Group. Dexmedetomidine vs midazolam for sedation of critically ill patients: a randomized trial. JAMA. 2009 Feb 4;301(5):489-99. doi: 10.1001/jama.2009.56. Epub 2009 Feb 2. PMID 19188334
- [Background] Pandharipande PP, Sanders RD, Girard TD, McGrane S, Thompson JL, Shintani AK, Herr DL, Maze M, Ely EW; MENDS investigators. Effect of dexmedetomidine versus lorazepam on outcome in patients with sepsis: an a priori-designed analysis of the MENDS randomized controlled trial. Crit Care. 2010;14(2):R38. doi: 10.1186/cc8916. Epub 2010 Mar 16. PMID 20233428
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Skrobik Y, Duprey MS, Hill NS, Devlin JW. Low-Dose Nocturnal Dexmedetomidine Prevents ICU Delirium. A Randomized, Placebo-controlled Trial. Am J Respir Crit Care Med. 2018 May 1;197(9):1147-1156. doi: 10.1164/rccm.201710-1995OC. PMID 29498534
- [Background] Reade MC, Eastwood GM, Bellomo R, Bailey M, Bersten A, Cheung B, Davies A, Delaney A, Ghosh A, van Haren F, Harley N, Knight D, McGuiness S, Mulder J, O'Donoghue S, Simpson N, Young P; DahLIA Investigators; Australian and New Zealand Intensive Care Society Clinical Trials Group. Effect of Dexmedetomidine Added to Standard Care on Ventilator-Free Time in Patients With Agitated Delirium: A Randomized Clinical Trial. JAMA. 2016 Apr 12;315(14):1460-8. doi: 10.1001/jama.2016.2707. PMID 26975647
- [Background] Burry L, Hutton B, Williamson DR, Mehta S, Adhikari NK, Cheng W, Ely EW, Egerod I, Fergusson DA, Rose L. Pharmacological interventions for the treatment of delirium in critically ill adults. Cochrane Database Syst Rev. 2019 Sep 3;9(9):CD011749. doi: 10.1002/14651858.CD011749.pub2. PMID 31479532
- [Background] Huupponen E, Maksimow A, Lapinlampi P, Sarkela M, Saastamoinen A, Snapir A, Scheinin H, Scheinin M, Merilainen P, Himanen SL, Jaaskelainen S. Electroencephalogram spindle activity during dexmedetomidine sedation and physiological sleep. Acta Anaesthesiol Scand. 2008 Feb;52(2):289-94. doi: 10.1111/j.1399-6576.2007.01537.x. Epub 2007 Nov 14. PMID 18005372
- [Background] Akeju O, Brown EN. Neural oscillations demonstrate that general anesthesia and sedative states are neurophysiologically distinct from sleep. Curr Opin Neurobiol. 2017 Jun;44:178-185. doi: 10.1016/j.conb.2017.04.011. Epub 2017 May 22. PMID 28544930
- [Background] Akeju O, Hobbs LE, Gao L, Burns SM, Pavone KJ, Plummer GS, Walsh EC, Houle TT, Kim SE, Bianchi MT, Ellenbogen JM, Brown EN. Dexmedetomidine promotes biomimetic non-rapid eye movement stage 3 sleep in humans: A pilot study. Clin Neurophysiol. 2018 Jan;129(1):69-78. doi: 10.1016/j.clinph.2017.10.005. Epub 2017 Oct 20. PMID 29154132
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Jorm AF. A short form of the Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE): development and cross-validation. Psychol Med. 1994 Feb;24(1):145-53. doi: 10.1017/s003329170002691x. PMID 8208879
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Inouye SK, Kosar CM, Tommet D, Schmitt EM, Puelle MR, Saczynski JS, Marcantonio ER, Jones RN. The CAM-S: development and validation of a new scoring system for delirium severity in 2 cohorts. Ann Intern Med. 2014 Apr 15;160(8):526-533. doi: 10.7326/M13-1927. PMID 24733193
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Rood P, Frenzel T, Verhage R, Bonn M, van der Hoeven H, Pickkers P, van den Boogaard M. Development and daily use of a numeric rating score to assess sleep quality in ICU patients. J Crit Care. 2019 Aug;52:68-74. doi: 10.1016/j.jcrc.2019.04.009. Epub 2019 Apr 6. PMID 30981928
- [Background] Gelinas C, Johnston C. Pain assessment in the critically ill ventilated adult: validation of the Critical-Care Pain Observation Tool and physiologic indicators. Clin J Pain. 2007 Jul-Aug;23(6):497-505. doi: 10.1097/AJP.0b013e31806a23fb. PMID 17575489
- [Background] Ferreira FL, Bota DP, Bross A, Melot C, Vincent JL. Serial evaluation of the SOFA score to predict outcome in critically ill patients. JAMA. 2001 Oct 10;286(14):1754-8. doi: 10.1001/jama.286.14.1754. PMID 11594901
- [Background] Woods SP, Delis DC, Scott JC, Kramer JH, Holdnack JA. The California Verbal Learning Test--second edition: test-retest reliability, practice effects, and reliable change indices for the standard and alternate forms. Arch Clin Neuropsychol. 2006 Aug;21(5):413-20. doi: 10.1016/j.acn.2006.06.002. Epub 2006 Jul 14. PMID 16843636
- [Background] Erdodi LA, Abeare CA, Lichtenstein JD, Tyson BT, Kucharski B, Zuccato BG, Roth RM. Wechsler Adult Intelligence Scale-Fourth Edition (WAIS-IV) processing speed scores as measures of noncredible responding: The third generation of embedded performance validity indicators. Psychol Assess. 2017 Feb;29(2):148-157. doi: 10.1037/pas0000319. Epub 2016 Apr 28. PMID 27124099
- [Background] Lee JH, Cheng R, Graff-Radford N, Foroud T, Mayeux R; National Institute on Aging Late-Onset Alzheimer's Disease Family Study Group. Analyses of the National Institute on Aging Late-Onset Alzheimer's Disease Family Study: implication of additional loci. Arch Neurol. 2008 Nov;65(11):1518-26. doi: 10.1001/archneur.65.11.1518. PMID 19001172
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Andresen EM, Malmgren JA, Carter WB, Patrick DL. Screening for depression in well older adults: evaluation of a short form of the CES-D (Center for Epidemiologic Studies Depression Scale). Am J Prev Med. 1994 Mar-Apr;10(2):77-84. PMID 8037935
- [Background] Djaiani G, Silverton N, Fedorko L, Carroll J, Styra R, Rao V, Katznelson R. Dexmedetomidine versus Propofol Sedation Reduces Delirium after Cardiac Surgery: A Randomized Controlled Trial. Anesthesiology. 2016 Feb;124(2):362-8. doi: 10.1097/ALN.0000000000000951. PMID 26575144
- [Background] Sun H, Ganglberger W, Panneerselvam E, Leone MJ, Quadri SA, Goparaju B, Tesh RA, Akeju O, Thomas RJ, Westover MB. Sleep staging from electrocardiography and respiration with deep learning. Sleep. 2020 Jul 13;43(7):zsz306. doi: 10.1093/sleep/zsz306. PMID 31863111
- [Background] Banks S, Dinges DF. Behavioral and physiological consequences of sleep restriction. J Clin Sleep Med. 2007 Aug 15;3(5):519-28. PMID 17803017
- [Background] Duff K. Evidence-based indicators of neuropsychological change in the individual patient: relevant concepts and methods. Arch Clin Neuropsychol. 2012 May;27(3):248-61. doi: 10.1093/arclin/acr120. Epub 2012 Feb 29. PMID 22382384
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Derived] Leone MJ, Dashti HS, Coughlin B, Tesh RA, Quadri SA, Bucklin AA, Adra N, Krishnamurthy PV, Ye EM, Hemmige A, Rajan S, Panneerselvam E, Higgins J, Ayub MA, Ganglberger W, Paixao L, Houle TT, Thompson BT, Johnson-Akeju O, Saxena R, Kimchi E, Cash SS, Thomas RJ, Westover MB. Sound and light levels in intensive care units in a large urban hospital in the United States. Chronobiol Int. 2023 Jun 3;40(6):759-768. doi: 10.1080/07420528.2023.2207647. Epub 2023 May 5. PMID 37144470
- See also: Airgo™ [Internet]. Airgo™. [cited 2022 Jul 8]. Available from: https://www.myairgo.com — https://www.myairgo.com
- See also: Heller LJ, Skinner CS, Tomiyama AJ, Epel ES, Hall PA, Allan J, et al. Trail-Making Test. In: Gellman MD, Turner JR, editors. Encyclopedia of Behavioral Medicine [Internet]. New York, NY: Springer New York; 2013 [cited 2022 Jul 8]. p. 1986-7. — http://link.springer.com/10.1007/978-1-4419-1005-9_1538
- See also: Brandt J, Spencer M, Folstein M. The Telephone Interview for Cognitive Status. Neuropsychiatry, Neuropsychology and Behavioral Neurology. 1988 Jan 1;1(2):111-7. — https://pure.johnshopkins.edu/en/publications/the-telephone-interview-for-cognitive-status-3
- See also: Fish J. Rankin Scale. In: Kreutzer JS, DeLuca J, Caplan B, editors. Encyclopedia of Clinical Neuropsychology [Internet]. New York, NY: Springer New York; 2011 [cited 2022 Jul 8]. p. 2110-2. — http://link.springer.com/10.1007/978-0-387-79948-3_1829
- See also: Gierveld JDJ, Tilburg TV. A 6-Item Scale for Overall, Emotional, and Social Loneliness: Confirmatory Tests on Survey Data. Res Aging. 2006 Sep;28(5):582-98. — https://core.ac.uk/download/pdf/18453043.pdf
- See also: Computing Comorbidity Scores (Charlson Comorbidity Index) — https://cran.r-project.org/web/packages/comorbidity/comorbidity.pdf

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT03355053/SAP_000.pdf